CLINICAL TRIAL: NCT05743387
Title: Community-based, eHealth Supported Type 2 Diabetes Care by Lay Village Health Workers in Rural Lesotho Protocol for a Cluster-randomized Trial Within the ComBaCaL Cohort Study (ComBaCaL T2D TwiC)
Brief Title: Community-based, eHealth Supported Type 2 Diabetes Care by Lay Village Health Workers in Rural Lesotho
Acronym: ComBaCaL T2D
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss Agency for Development and Cooperation (SDC) (Unknown); World Diabetes Foundation (WDF) (Unknown); SolidarMed (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AO_2022-00077; am23Labhardt
Record Dates: First submitted 2023-02-14; First posted 2023-02-24 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes Mellitus (T2D)
Keywords: Community-Based Chronic Disease Care Lesotho (ComBaCaL) cohort study; low- and middle-income countries (LMICs); lay healthcare worker (LHW); chronic care village health worker (CC-VHW); chronic care nurse (CC nurse); non-communicable disease (NCD); blood glucose (BG); cardiovascular disease risk factor (CVDRF); glycated haemoglobin (HbA1c); Lesotho Ministry of Health (MoH) Village Health Worker Program; first-line antidiabetics; first-line lipid-lowering treatment
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Noncommunicable Diseases

STUDY DESIGN:
Intervention Model Description: Cluster-randomized controlled trial nested within the ComBaCaL cohort study following a trial within cohort (TwiC) approach. 50% of the villages being part of the overarching ComBaCaL cohort will be randomized stratified by district and access to health facility to receive the intervention.
Who Masked: Outcomes Assessor
Masking Description: Participants are not blinded to the intervention due to the nature of the intervention. Due to the cluster level randomization and TwiCs approach participants are blinded to the allocation (i.e. participants in the control villages are not aware of the intervention being implemented in the intervention villages). The main outcome and the safety endpoints are assessed by an independent study physician blinded to the allocation. The statistician and data managers cannot be blinded to the allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention villages (Active Comparator): In the intervention villages, CC-VHWs will offer
  * a T2D care package including lifestyle counselling, firstline antidiabetic (metformin) and lipid-lowering (statin) treatment for uncomplicated T2D and treatment support and regular check-ups for complicated T2D at village-level according to clinical algorithms based on international guidelines for primary healthcare management of T2D and the updated Lesotho Standard Treatment Guidelines.
  * Direct guidance for treatment initiation, drug prescription, counselling and monitoring will be provided via the ComBaCaL app.
  * In case of complicated disease (i.e. if treatment targets are not reached with metformin alone), unclear diagnosis, relevant comorbidities or presence of clinical alarm signs or symptoms, participants will be referred to the closest health facility for further management.
  Interventions: Other: T2D care package
- Control villages (Active Comparator): In control villages, CC-VHWs will refer participants to the responsible health facility for therapeutic management after enrolment and baseline assessment.
  Interventions: Other: Referral to the responsible health facility

INTERVENTIONS:
Other: T2D care package — T2D care package including lifestyle counselling, firstline antidiabetic (metformin) and lipid-lowering (statin) treatment for uncomplicated T2D and treatment support and regular check-ups for complicated T2D at village-level. Guidance will be provided via the ComBaCaL app. In case of complicated disease referral to the closest health facility for further management.
  Arms: Intervention villages
Other: Referral to the responsible health facility — CC-VHWs will refer participants to the responsible health facility for therapeutic management. The ComBaCaL app supports clinical decision making and documentation for screening, diagnosis and referral, but not prescription/provision and monitoring of antidiabetic or lipid-lowering medication for uncomplicated T2D patients or treatment support for complicated T2D patients.
  Arms: Control villages

SUMMARY:
This cluster-randomized intervention is embedded in the ComBaCaL (Community-Based Chronic disease care Lesotho) cohort study (EKNZ ID AO_2022-00058, clinicaltrials.gov ID NCT05596773, Lesotho NH-REC ID 210-2022), a platform for the investigation of chronic diseases and their management in rural Lesotho that is maintained by local lay chronic care village health workers (CC-VHWs).

The overall objective of the ComBaCaL cohort study and nested TwiCs is to assess the impact of eHealthsupported, lay-led chronic disease control measures in rural Lesotho.

In this T2D TwiC, the effect, safety and feasibility of a community-based T2D care package (which includes the offer of first-line oral antidiabetic and lipid-lowering treatment for uncomplicated T2D by lay CC-VHWs in comparison to facility-based care after community-based screening and diagnosis) will be evaluated.

DETAILED DESCRIPTION:
Globally, 9.3% of the adult population or 436 million individuals were estimated to be living with diabetes in 2019. Until 2045 this number is expected to increase by more than 50% to over 700 million. Four out of five people affected by diabetes are currently living in low- and middle-income countries (LMICs). Over 90% of all diabetes cases are due to type 2 diabetes (T2D) which is also the main driver of the projected increase in overall diabetes cases. The increase in T2D prevalence is caused by ageing populations and changing lifestyles with decreasing levels of physical activity and higher caloric diets and associated obesity.

This cluster-randomized intervention is embedded in the ComBaCaL (Community-Based Chronic disease care Lesotho) cohort study (EKNZ ID AO_2022-00058, clinicaltrials.gov ID NCT05596773, Lesotho NH-REC ID 210-2022), a platform for the investigation of chronic diseases and their management in rural Lesotho that is maintained by local lay chronic care village health workers (CC-VHWs).

In this trial, using the Trials within Cohorts (TwiCs) approach, it will be analyzed whether an LHW-led model could be capacitated to safely and effectively provide first-line management (including oral antidiabetic, lipid-lowering treatment and lifestyle counselling) at community-level.

In villages randomized to the intervention arm, lay Chronic Care Village Health Workers (CCVHWs) operating within the existing Ministry of Health (MoH) village health worker system will be capacitated to screen for and diagnose T2D, to provide lifestyle counselling, to prescribe and to monitor first-line antidiabetic and lipid-lowering treatment for uncomplicated T2D and to provide treatment support for complicated T2D, supported by a tailored clinical decision support application (ComBaCaL app) in their villages.

The control group consists of people diagnosed with T2D living in villages that are also part of the ComBaCaL cohort but not sampled for the intervention (control villages), where CC-VHWs will only screen for and diagnose T2D with subsequent standardized counselling and referral to the closest health facility if T2D is present, but no village-based prescriptions. The overall objective of the ComBaCaL cohort study and nested TwiCs is to assess the impact of eHealthsupported, lay-led chronic disease control measures in rural Lesotho.

ELIGIBILITY:
Inclusion Criteria:

* Participant of the ComBaCaL cohort study (signed informed consent available)
* Living with T2D, defined as reporting intake of antidiabetic medication or being newly diagnosed during screening via standard diagnostic algorithm

Exclusion Criteria:

* Known type 1 diabetes mellitus
* Reported pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2023-05-13 (Actual); Primary Completion 2025-03-23 (Actual); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Mean HbA1c (in percent) | 12 months after enrolment
  Mean HbA1c (in percent)

SECONDARY OUTCOMES:
Change in 10-year CVD risk estimated | 6 and 12 months after enrolment
  Change in 10-year CVD risk estimated using the World Health Organization (WHO) CVD risk prediction tool
Mean HbA1c (in percent) | 6 months after enrolment
  Mean HbA1c (in percent)
Change in mean fasting blood glucose (FBG) (mmol/l) | 6 and 12 months after enrolment
  Change in mean fasting blood glucose (FBG) (mmol/l)
Change in proportion of participants with an HbA1c below 8% | 6 and 12 months after enrolment
  Change in proportion of participants with an HbA1c below 8%
Change in proportion of participants with an FBG below 7 mmol/l | 6 and 12 months after enrolment
  Change in proportion of participants with an FBG below 7 mmol/l
Change in number of CVD risk factors | 6 and 12 months after enrolment
  Change in number of CVD risk factors (such as smoking status, BMI, abdominal circumference, blood lipid status, blood pressure, dietary habits and physical activity)
Linkage to care: Change in proportion of participants not taking treatment at enrolment who have initiated pharmacological antidiabetic treatment | 6 and 12 months after enrolment
  Change in proportion of participants not taking treatment at enrolment who have initiated pharmacological antidiabetic treatment
Engagement in care: Change in proportion of participants who are engaged in care | 6 and 12 months after enrolment
  Change in proportion of participants who are engaged in care, defined as reporting intake of antidiabetic medication as per prescription of a healthcare provider or reaching treatment targets without intake of medication
Change in self-reported adherence to antidiabetic medication | 6 and 12 months after enrolment
  Change in self-reported adherence to antidiabetic medication
Occurrence of Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESIs) | within 6 and 12 months after enrolment
  Occurrence of Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESIs)

OTHER OUTCOMES:
Number of consultations (at a health facility and with the CC-VHW) | within 6 and 12 months after enrolment
  Number of consultations at a health facility and with the CC-VHW
Trajectory of participants between facility-based and community-based care in the intervention villages | during the study period (up to 12 months)
  Trajectory of participants between facility-based and community-based care in the intervention villages (i.e. number of participants accepting community-based care at baseline, number of people switching to facility-based care and back to community-based care
Proportion of participants with T2D who stop drug treatment or interrupt drug treatment for more than three weeks or require a switch of drug treatment due to (perceived) adverse events (AEs) | within 6 and 12 months after enrolment
  Proportion of participants with T2D who stop drug treatment or interrupt drug treatment for more than three weeks or require a switch of drug treatment due to (perceived) adverse events (AEs)
Change in proportion of participants who are reaching treatment targets (FBG <7 mmol/l) and are reporting no intake of antidiabetic medication in the two weeks prior to assessment | 6 and 12 months after enrolment
  Change in proportion of participants who are reaching treatment targets (FBG <7 mmol/l) and are reporting no intake of antidiabetic medication in the two weeks prior to assessment
Change in proportion of participants accessing lipid-lowering medication | 6 and 12 months after enrolment
  Change in proportion of participants accessing lipid-lowering medication
Change in health system costs for the management of participants condition | within 6 and 12 months after diagnosis
  Change in health system costs for the management of participants condition
Change in individual costs for participants for the management of their condition | within 6 and 12 months after diagnosis
  Change in individual costs for participants for the management of their condition
Change in10-year CVD risk estimated using the Globorisk score | 6 and 12 months after enrolment
  Change in10-year CVD risk estimated using the Globorisk score, a cardiovascular disease risk score that predicts risk of heart attack or stroke in healthy individuals for all countries in the world. It uses information on a person's country of residence, age, sex, smoking, diabetes, blood pressure and cholesterol to predict the chance that they would have a heart attack or stroke in the next 10 years.
Change in10-year CVD risk estimated using the Framingham Risk Score | 6 and 12 months after enrolment
  Change in10-year CVD risk estimated using the Framingham Risk Score, a sex-specific algorithm used to estimate the 10-year cardiovascular risk of an individual. The Framingham Risk Score was first developed based on data obtained from the Framingham Heart Study.
Quality of life (QOL) using the EQ-5D-5L instrument | 12 months after enrolment
  The EQ-5D-5L is a self-assessed, health related, quality of life questionnaire. The scale measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The QOL scores are summed so that a higher score indicates higher quality of life.
Health beliefs using the Beliefs about Medicines Questionnaire (BMQ) adapted for people living with T2D | 12 months after enrolment
  The BMQl comprises two 4-item factors assessing beliefs that medicines are harmful, addictive, poisons which should not be taken continuously and that medicines are overused by doctors.The items are scored on a 5 point Likert scale with scores ranging from 4 to 20.
Diabetes distress using the five item version of the "Problem Areas in Diabetes" (PAID-5) scale Problem Areas in Diabetes Scale-Five-item Short Form | 12 months after enrolment
  Problem Areas in Diabetes Scale-Five-item Short Form. Total scores on the PAID-5 can range from 0 to 20, with higher scores suggesting greater diabetes-related emotional distress.
Change in dosage of antidiabetic medications prescribed by CC-VHWs or healthcare professionals | 6 and 12 months after enrolment
  Change in dosage of antidiabetic medications prescribed by CC-VHWs or healthcare professionals
Change in dosage of lipid-lowering medications prescribed by CC-VHWs or healthcare professionals | 6 and 12 months after enrolment
  Change in dosage of lipid-lowering medications prescribed by CC-VHWs or healthcare professionals

CONTACTS AND LOCATIONS:
Overall Officials: Niklaus Labhardt, Prof., Principal Investigator — Division of Clinical Epidemiology, University Hospital Basel; Alain Amstutz, MD, Principal Investigator — Division of Clinical Epidemiology, University Hospital Basel, University of Basel
Locations (2):
- SolidarMed Lesotho, Maseru, Lesotho
- University of Basel, Division of Clinical Epidemiology, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
* An anonymized key dataset necessary for reproducing the primary and key secondary endpoints will be made freely available in an appropriate repository, such as zenodo.org, alongside the publication of the study results. Besides removal of variables not required for key analysis, we will remove participant identifier, study site and exact date information. Requests for access to more detailed data may be made to the corresponding author by submitting a proposal, which will be reviewed by the trial consortium.
  * The statistical report for the primary and key secondary endpoints and the code to produce it will be published together with the data set.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: • Within 3 months after publication of primary results
Access Criteria: • Open access

REFERENCES:
- [Derived] Gerber F, Gupta R, Lejone TI, Tahirsylaj T, Lee T, Kohler M, Haldemann MI, Raber F, Chitja M, Manthabiseng M, Khomolishoele M, Mota M, Bane M, Sematle PM, Makabateng R, Mphunyane M, Phaaroe S, Basler D, Kindler K, Seelig E, Briel M, Chammartin F, Labhardt ND, Amstutz A. Community-based type 2 diabetes care by lay village health workers in rural Lesotho: protocol for a cluster-randomized trial within the ComBaCaL cohort study (ComBaCaL T2D TwiC). Trials. 2023 Oct 24;24(1):688. doi: 10.1186/s13063-023-07729-8. PMID 37875943

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Protocol (2023-02-03): https://cdn.clinicaltrials.gov/large-docs/87/NCT05743387/Prot_SAP_000.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan (2024-11-21): https://cdn.clinicaltrials.gov/large-docs/87/NCT05743387/SAP_001.pdf